CLINICAL TRIAL: NCT00416299
Title: Observational Cohort Study on the Prognostic Value of New Cardiac Biomarkers in Elderly Patients Undergoing Cardiac Surgery
Brief Title: Prognostic Value of New Cardiac Biomarkers in Elderly Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Other Study IDs: KliLuNTproBNP
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Cardiac Surgery
Keywords: Cardiac biomarker; cardiac surgery; elderly; postoperative complications; Patients aged 75 years or older undergoing cardiac surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the use of new cardiac biomarker for the prediction of in-hospital cardiovascular complications in elderly patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Plasma N-terminal pro-brain natriuretic peptide (NT-proBNP, cardiac troponin T (cTnT), pregnancy-associated plasma protein A (PAPP-A), ischemia-modified albumin (IMA), myeloperoxidase (MPO), metalloproteinase (MMP) soluble CD 40 ligand (sCD40L), and inflammatory cytokine levels will be measured in 100 elderly patients undergoing elective cardiac surgery with cardiopulmonary bypass before induction of anesthesia and 12 h, 24 h, and 48 h after surgery. Optimum discriminators for prediction of postoperative cardiovascular complications wil be determined by the use of receiver operating characteristics (ROC) curves analyses.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 75 years or older undergoing elective cardiac surgery with CPB

Exclusion Criteria:

* positive cardiac troponin T test within the week before surgery
* patients undergoing emergent procedures
* patients with preoperative mechanical cardiac support
* patients undergoing hemodialysis

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan W. Suttner, MD, Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Klinikum Ludwigshafen, Ludwigshafen, Germany